CLINICAL TRIAL: NCT06615544
Title: Clinical Evaluation of a New Dual-cure Universal Adhesive for Indirect Restorative Treatment
Brief Title: Clinical Evaluation of a New Dual-cure Universal Adhesive
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ivoclar Vivadent AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OTCS187092274
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Results first posted 2025-08-19 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-08

CONDITIONS: Class I Dental Restorations; Class II Dental Restorations; Insufficient Dental Restoration; Caries, Dental
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- New dual-cure adhesive (Experimental): The newly developed dual-cure adhesive will be used for the placement of indirect restorations.
  Interventions: Device: Placement of indirect dental restoration

INTERVENTIONS:
Device: Placement of indirect dental restoration — The newly developed dual-cure adhesive will be used for the placement of indirect restorations.

SUMMARY:
The overall aim of this study is to evaluate the clinical performance and safety of the new dental dual-cure adhesive for luting indirect ceramic restorations (inlays and onlays). The primary aim is to determine the rate of postoperative hypersensitivity occurrence after using the new adhesive for the placement of indirect restorations. The secondary objective of this study is to assess the long-term clinical performance of the new adhesive in terms of marginal quality, retention/fracture rate of the ceramic restorations, and vitality/fracture rate of the restored teeth.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years
* Informed consent signed and understood by the subject
* Indication for indirect restorations (inlay, onlay) in molar or premolar
* The occlusal area of the restoration must cover at least 1/3 of the occlusal area of the tooth.
* visual analogue scale (VAS)<4 (0=no pain, 10=maximum conceivable pain)
* Max. 2 restorations per participant in different quadrants.
* Vital tooth
* Healthy periodontium, no active periodontitis
* Contact with adjacent teeth (at least at one side) and opposing teeth present with at least one contact point.
* Sufficient language skills

Exclusion Criteria:

* Insufficient isolation
* Participants with a proven allergy to one of the ingredients of the materials used
* Participants with proven allergy to local anaesthetics
* High caries activity/ poor oral hygiene
* Participants with severe systemic diseases
* Pregnancy
* Tooth with irreversible pulpitis
* Indication for direct pulp capping
* Bleaching of teeth within the last 14 days
* Usage of peroxide-based disinfectants within the last 14 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2031-04 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Ivoclar Vivadent AG, Schaan, Liechtenstein, Liechtenstein

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Restorations
Period: Overall Study
Arm/Group | New dual-cure adhesive
Started | 45; 48 Restorations
Completed | 45; 47 Restorations
Not Completed | 0; 1 Restorations

BASELINE CHARACTERISTICS:
Units Other Than Participants: Restorations
Arm/Group | New dual-cure adhesive
Number analyzed (Participants) | 45
Number analyzed (Restorations) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Hypersensitivity
Description: will be assessed according to FDI criteria (grade 1-5, lower scores mean a better outcome)
Time Frame: 1 month
Population: One patient was not able to visit 1-month recall (no-show)
Measure: Number; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | New dual-cure adhesive
Number analyzed (Participants) | 44
Number analyzed (Restorations) | 46
Restorations
  FDI Score 1 | 46
  FDI Score 2-5 | 0

2. Secondary Outcome: Fracture Rate
Description: will be assessed according to FDI criteria (grade 1-5, lower scores mean a better outcome)
Time Frame: 5 years
Reporting Status: Not Posted

3. Secondary Outcome: Marginal Quality
Description: will be assessed according to FDI criteria (grade 1-5, lower scores mean a better outcome)
Time Frame: 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1-Month
Arm/Group | New dual-cure adhesive
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 3/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | New dual-cure adhesive (N=45)
Unrealated: Cementation Mistake (General disorders) | 1 — Restoration was removed before Baseline and a new one with a standard workflow was placed. Cementation mistake is unrelated to the test product
Unrealated: Cementation Mistake (General disorders) | 2 — Cementation mistake of a restoration occured, which is unrelated to the test product. Restorations were not replaced and patients are symptom-free.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT06615544/Prot_SAP_001.pdf